CLINICAL TRIAL: NCT00974402
Title: Psychotherapy Treatment of Deployment-related PTSD in Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); 59th Medical Wing (U.S. Federal Agency); South Texas Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20090194H; BAMC C.2009.022 (Other: Brooke Army Medical Center Institutional Review Board); W81XWH-08-2-0109 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Post-Traumatic Stress Disorders; Stress Disorders; Combat Disorders
Keywords: Active duty; Afghanistan; Anger; Anxiety; Avoidance; BAMC; Brooke Army Medical Center; Cognitive Behavioral Therapy; Combat; Combat Disorder; Coping; Counseling; Counselor; Deployment; Depression; Exposure; Fear; Feeling alone; Flashbacks; Guard; Guilt; Hospitalization; Iraq; Mental Health; Military; Military member; Military personnel; Neuroses; Nightmares; OEF; OIF; Prolonged Exposure Therapy; Psychiatric; Psychiatric medication; Psychological distress; Psychotherapy; Reserve; Retired; Sadness; Separated; Sleeplessness; Soldier; Stress; Stress disorder; Stress management; STRONG STAR; Suicidal; Suicide; Therapy; Trauma; Traumatic Event; Trouble Sleeping; Veteran; Veterans; War; WHMC; Wilford Hall Medical Center; PTSD; Posttraumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Combat Disorders; Anxiety Disorders; Depression; Psychological Well-Being; Neurotic Disorders; Sleep Initiation and Maintenance Disorders; Suicide; Wounds and Injuries; Parasomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with PTSD Symptoms (Experimental): Patients with Post-Traumatic Stress Disorder (PTSD) symptoms willing to undergo Cognitive Behavioral Therapy in a primary care setting.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The study investigators have developed a 4-session PTSD treatment plan including a behavioral health consultants (BHC) manual and a patient guide for use in primary care. Therapists will be psychologists who are functioning as behavioral health consultants (BHC) in an integrated primary care clinic. The study will adapt intervention methods for use in the time-constrained primary care environment from Cognitive Behavioral Therapy(ies) that have proven effective for PTSD in specialty mental health care settings. Study participants will receive four 30-minute treatment sessions over six weeks.
  Other Names: brief cognitive-behavioral therapy (CBT)

SUMMARY:
The purpose of this study is to evaluate Cognitive-behavioral therapy (CBT) for deployment-related post-traumatic stress disorder (PTSD) that can be used by behavioral health consultants working with Service Members in the primary care clinic. CBT is a well-researched, very effective individual (one-to-one) treatment that is designed to help people to directly deal with traumatic events they have suffered in the past, including combat. Many Service Members prefer to see behavioral health providers in primary care rather than the mental health clinic. The researchers hope to learn if a brief treatment for PTSD in primary care can be just as useful as more traditional treatment given in the mental health clinic. This study will enroll approximately 45 participants overall; with approximately 30 participants at Wilford Hall Medical Center or Brooke Army Medical Center, and 15 participants to be enrolled at the South Texas Veterans Health Care System over a period of one year.

ELIGIBILITY:
Inclusion Criteria:

* The target population for the study is active duty, reserve, guard, separated, or retired OIF/OEF veterans (minimum age 18 and English speaking) in the primary care population who are symptomatic for deployment-related PTSD and interested in treatment.
* Symptomatic for PTSD will be defined as a minimum score of 32 on the PTSD CheckList - Military (PCL-M).

Exclusion Criteria:

* The exclusion criteria are those that would normally apply for standard of care behavioral health consultation in an integrated primary care clinic.
* These exclusion criteria are moderate to severe suicide risk, current alcohol dependence, psychotic disorder, significant dissociative disorder, and severe brain injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
PTSD symptomatology | Baseline, post-treatment, 6-month and 12-month
  PTSD symptoms as assessed by an evaluator-administered interview (PTSD Symptom Scale Interview - PSSI) and self-report form (PTSD Checklist - Military Version - PCL-M).

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Peterson, PhD, Study Chair — University of Texas Health Science Center San Antonio (UTHSCSA), STRONG STAR Consortium Director; Jeffrey Cigrang, Lt Col, Principal Investigator — U.S. Air Force, 5MDG, Minot Air Force Base; Lisa Kearney, PhD, Principal Investigator — South Texas Veterans Health Care System (STVHCS); Diana Dolan, Capt, Principal Investigator — U.S. Air Force, Wilford Hall Medical Center (WHMC); Laura Avila, PhD, Principal Investigator — Brooke Army Medical Center
Locations (3):
- United States (3):
  - South Texas Veterans Health Care System (STVHCS), San Antonio, Texas
  - Brooke Army Medical Center (BAMC), San Antonio, Texas
  - Wilford Hall Medical Center, San Antonio, Texas

REFERENCES:
- See also: Related Info — http://www.strongstar.org